CLINICAL TRIAL: NCT01423032
Title: Bendamustine Versus Fludarabine as 2nd-line Treatment in Chronic Lymphocytic Leukemia, Stage BINET B+C / RAI II-IV
Brief Title: Bendamustine Versus Fludarabine in Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: WiSP Wissenschaftlicher Service Pharma GmbH (Other)
Collaborators: Klinikum Leverkusen gGmbH (Unknown); ribosepharm GmbH (Unknown); Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WISP_RI05
Record Dates: First submitted 2011-08-19; First posted 2011-08-25 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: relapsed
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — Bendamustine Hydrochloride; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bendamustine (Experimental)
  Interventions: Drug: bendamustine
- Fludarabine (Active Comparator)
  Interventions: Drug: Fludarabine

INTERVENTIONS:
Drug: bendamustine — 100 mg/m² iv, day 1+2, q4w
  Arms: Bendamustine
Drug: Fludarabine — 25 mg/m² iv, days 1-5, q4w
  Arms: Fludarabine

SUMMARY:
Bendamustine demonstrated clinical activity in pre-treated hematological malignancies due to its unique mechanism of action distinct from standard alkylating agents. This study assesses its efficacy in patients with chronic lymphocytic leukemia pre-treated with an alkylator, in comparison to fludarabine.

Patients with relapsed chronic lymphocytic leukemia requiring treatment after one previous systemic regimen (usually chlorambucil-based) are randomized to either receive bendamustine 100 mg/m² on days 1 and 2 of a 4-week cycle, or standard fludarabine treatment consisting of 25 mg/m² on days 1 to 5 every four weeks. The primary objective was to achieve non-inferior progression-free survival with bendamustine.

ELIGIBILITY:
Inclusion Criteria:

* histologically or immunologically confirmed chronic B-cell leukemia
* refractory (i.e. no response or progression during initial chemotherapy) or relapsed situation after first-line treatment regimen
* disease stage II-IV according to Rai or B/C according to Binet staging system, respectively
* Eastern Cooperative Oncology Group (ECOG) performance status of 3 or better
* negative pregnancy test/ adequate method of contraception

Exclusion Criteria:

* T-CLL, PLL (prolymphocytic leukemia)
* presence of Richter's transformation
* first-line treatment containing either fludarabine or bendamustine
* acute infections or distinctly reduced organ function precluding the application of chemotherapy, as for pulmonary, heart, liver (total bilirubin > 5mg/dl), renal system (creatinine > 2 mg/dl), or metabolic disorders
* secondary malignancy (except for curative treated basal cell carcinoma or cervical cancer)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2001-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
progression-free survival | the patients were followed on average for 36 months
  individual time-frame up to max. follow-up (Kaplan-Meier estimation)

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Niederle, Prof, MD, Study Chair — Med. Klinik III, Klinikum Leverkusen gGmbH, Germany
Locations (1):
- Prof. Dr. Norbert Niederle, Leverkusen, North Rhine-Westphalia, Germany